CLINICAL TRIAL: NCT00329368
Title: A Phase I Study of EC90 With GPI-0100 Adjuvant Followed by EC17 With Cytokines (Interleukin-2 [IL-2] and Interferon-alpha [IFN-alpha]) in Patients With Refractory or Metastatic Cancer
Brief Title: Safety and Tolerability Study of FolateImmune in Combination With Cytokines in Patients With Refractory or Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Endocyte (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC-FI-003
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Cancer
Keywords: Cancer; Vaccine; Phase I; FolateImmune; Recurrent; Refractory; Experimental
MeSH Terms: conditions — Neoplasms; Recurrence | interventions — fluorescein isothiocyanate-keyhole limpet hemocyanin; GPI0100; Interleukin-2; aldesleukin; Interferon-alpha; Introns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: EC90 (KLH-FITC) — 1.2mg in combination with adjuvant GPI-0100 administered subcutaneously, weekly for 4 consecutive weeks during the first treatment cycle, weekly for 2 consecutive weeks during the second cycle and once for each additional cycle.
  Other Names: Keyhole limpet hemocyanin fluorescein
Biological: GPI-0100 — 3.0mg in combination with EC90 administered subcutaneously weekly for 4 consecutive weeks during the first treatment cycle, weekly for 2 consecutive weeks during the second cycle and once for each additional cycle.
  Other Names: Saponin-based adjuvant
Drug: EC17 (Folate-FITC) — 0.3mg/kg administered subcutaneously 5 days per week (Monday through Friday) for 4 consecutive weeks followed by 2 observation weeks for each cycle.
  Other Names: folate-fluorescein conjugate; folate-hapten conjugate
Drug: Interleukin-2 — Low dose (7-12 MIU) IL-2 administered subcutaneously three times per week (MWF) for 3 consecutive weeks during the first cycle, 4 consecutive weeks during cycle 2 and additional cycles
  Other Names: IL-2; Proleukin
Drug: Interferon-alpha — 3.0 MIU administered subcutaneously 3 times per week (MWF) for 3 consecutive weeks during the first cycle of treatment, then 3.0 MIU administered subcutaneously 3 times per week (MWF) for 4 weeks for cycle 2 and additional cycles.
  Other Names: IFN-alpha; Intron-A

SUMMARY:
This is a Phase 1b clinical trial to assess the safety and tolerability of vaccination with EC90 (KLH-FITC) and GPI-0100 (adjuvant) followed by treatment with EC17 (Folate-FITC) in combination with low-dose cytokines (IL-2 and IFN-alpha) in patients with metastatic or refractory cancer.

DETAILED DESCRIPTION:
Rationale: This is a Phase 1b, single-cohort study of FolateImmune in combination with low-doses of the cytokines Interleukin-2 (IL-2) and Interferon-alpha (IFN-alpha). FolateImmune treatment consists of subcutaneous vaccinations with EC90, a compound designed to elicit an immune response (antibodies) to a dye called fluorescein (FITC), in combination with GPI-0100 adjuvant (a drug intended to improve antibody production). Vaccination is followed by treatment with EC17, a drug made by linking folate (a vitamin) with FITC. Experimental evidence has shown that the folate vitamin receptor is over-expressed in many human cancers. It is expected that EC17 will attach to cancer cells through the folate vitamin receptor and that antibodies to FITC will recognize the cancer cell and mark it for destruction by the body's immune system. Two drugs, IL-2 and IFN-alpha, will be administered at low doses in combination with EC17 in order to boost the immune response.

Objectives:

* Evaluate the safety of administering EC90 vaccine with GPI-0100 adjuvant.
* Evaluate the safety of administering EC17 concurrent with IL-2 and IFN-alpha

ELIGIBILITY:
Inclusion Criteria:

* Have a histologically confirmed diagnosis of metastatic or refractory cancer for which there are no effective standard therapeutic options available, (Note: for patients accrued at Southern Illinois University, a diagnosis of renal (i.e., kidney) carcinoma is required.)
* Have signed an Institutional Review Board (IRB) approved informed consent form (ICF) prior to performing any study evaluation/procedures
* Be > or = 18 years of age and women must either be 1) not of childbearing potential or 2) have a negative serum pregnancy test within 7 days prior to commencing treatment. Patients are considered not of childbearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or they are postmenopausal (12 consecutive months of amenorrhea [lack of menstruation])
* (If applicable) Have completed prior cytotoxic chemotherapy, radiotherapy or immunotherapy or experimental therapy > or = 30 days prior to the study enrollment, and recovered form associated toxicities
* Have an Eastern Cooperative Oncology Group (ECOG) score of < or = 2, and an anticipated life expectancy of at least 6 months
* Have adequate hematologic function, as defined by an absolute or calculated neutrophil count > or = 1500/microL, platelet count > or = 100000/microL, lymphocyte count > or = 500/microL, and hemoglobin level > or = 10 g/dL. Patients may not receive prophylactic transfusion in order to qualify for trial eligibility
* Have adequate renal function, as defined by a documented serum creatinine of < or = 2.0mg/dL. Greater than "1+" proteinuria will require microscope evaluation and the results discussed with the medical monitor prior to patient enrollment; or if serum creatine is >2.0, patient must have an actual or calculated 24-hour creatinine clearance of >60mL/min and no obvious evidence of concurrent medullary cystic disease or obstructive uropathy
* Have adequate hepatic function, as defined by a total bilirubin level < or = 1.5 x upper limit of normal (ULN) and alkaline phosphatase, aspartate transaminase (AST), and alanine transaminase (ALT) levels < or = 2.5 x ULN. If alkaline phosphatase is outside of these parameters and is due to bone metastases (as verified by the assessment of isoenzymes), then the patient is eligible.

Exclusion Criteria:

* Have previously participated in a FolateImmune trial
* Have a history of severe hypersensitivity (grade 3 - 4 allergic reaction) to fluorescein or any drug, radiologic contrast agent, insect bite, food, cytokines, or any other agent; or have received fluorescein within 30 days of the study.
* Have medical conditions that preclude the use of IL-2 or IFN-alpha. These conditions include but are not limited to, diabetes mellitus with a history of progression to diabetic ketoacidosis, history of severe coagulation disorder, psoriasis, sarcoidosis, retinal hemorrhage, symptomatic pulmonary disease, heart failure (> or = New York Heart Association NYHA class II), or transplant requiring immunosuppressive therapy
* Be pregnant or breast-feeding
* Be currently receiving an experimental drug, or used an experimental device within 30 days of study entry
* Be currently undergoing chemotherapy, anticancer hormonal therapy, and/or therapy with immunosuppressant agents
* Have any concomitant malignancy with the exception of basal cell or squamous cell carcinoma of skin
* Have radiographically documented evidence of current brain metastases, a history of stem cell transplant, immunodeficiency, and/or a medical or psychiatric illness (that in the investigator's opinion, would prevent adequate compliance with study therapy or evaluation of the endpoints)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-09; Primary Completion 2007-12 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Safety | Initial dose of study therapy through 30 days post last dose of study therapy
Tolerability | Initial dose of study therapy through 30 days post last dose of study therapy
Anti-tumor Activity | From initial dose of study therapy to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Messmann, MD, MHS, BSc, Study Director — Endocyte
Locations (3):
- United States (3):
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Great Lakes Cancer Institute Breslin Cancer Center, Lansing, Michigan
  - The Methodist Hospital, Houston, Texas